CLINICAL TRIAL: NCT06792097
Title: The Role of Ga-68 Dolacga PET Scan in Patients With Hepatocellular Carcinoma Under Radiofrequency Ablation
Brief Title: Ga-68 Dolacga PET Scan in HCC Under RFA
Acronym: HCC; RFA
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202409045MIND
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma (HCC); Radiofrequency Ablation; PET Scan; Computed Tomography; Deep Learning
Keywords: Hepatocellular carcinoma; Radiofrequency ablation; Ga-68 Dolacga PET scan; Liver function; Neural network; Radiomics
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ga-68 Dolacga PET scan — Contrast Name: Nuclear Medicine Dolacga (Lyophilized product for the preparation of gallium Ga68 Dolacga injection).
  Active Ingredient, Dosage, Route: NOTA-Hexa lactoside (INER038), 40 micrograms, IV injection.
  PET Imaging Schedule: Before radiofrequency ablation therapy, one month after ablation therapy, and follow-up every three months thereafter.

SUMMARY:
This study aims to investigate the use of Ga-68 Dolacga PET scan technology to assess treatment response and liver function changes in patients of early-stage liver cancer receiving RFA. The main questions it aims to answer are:

1. How to assess treatment response and liver function changes in hepatocellular carcinoma patients undergo RFA via Ga-68 Dolacga PET scan?
2. Compared with computed tomography (CT) scans, how effective is Ga-68 Dolacga PET scan for treatment response assessment?
3. What is the correlation between Ga-68 Dolacga PET scan findings and patient treatment outcomes by tracking liver function and tumor recurrence after RFA?

Participants will:

1. Undergo Ga-68 Dolacga PET scans and computed tomography before and one month after RFA treatment, followed by monitoring every three months thereafter.
2. Total liver functional volume and residual liver functional volume are obtained from Ga-68 Dolacga PET scan

DETAILED DESCRIPTION:
This study aims to investigate the use of Ga-68 Dolacga PET scan technology to assess treatment response and liver function changes in patients of early-stage liver cancer receiving RFA. This study also compares the results of Ga-68 Dolacga PET scans with computed tomography (CT) scans and evaluate the correlation between Ga-68 Dolacga PET scan findings and patient treatment outcomes by tracking liver function and tumor recurrence after RFA.

This study adopts a prospective clinical trial design, enrolling patients with early-stage liver cancer and undergoing RFA treatment. Clinical data, laboratory results, serum, biopsy tissues for pathology and relevant imaging findings are collected for analysis. Participants undergo Ga-68 Dolacga PET scans and CT before and one month after RFA treatment, followed by monitoring every three months thereafter. Quantitative analysis utilizes region of interest techniques to measure standardized uptake values (SUV). Total liver functional volume and residual liver functional volume are obtained from Ga-68 Dolacga PET scan injection dose percentages and SUV values. Changes in liver storage capacity as determined by Ga-68 Dolacga PET scans are evaluated and correlated with traditional laboratory liver function tests and imaging evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatocellular carcinoma (BCLC stage 0 and stage A) eligible for radiofrequency ablation (RFA) treatment exhibit the following characteristics:

  1. A single liver tumor, ≤ 2 cm, classified as BCLC stage 0 (very early stage).
  2. Tumors ≤ 3 in number, each ≤ 3 cm, or a single tumor ≤ 5 cm, classified as BCLC stage A (early stage) liver cancer.
  3. ECOG performance status of 0.
  4. Age ≥ 18 years.

     Exclusion Criteria:
* Intermediate (BCLC B stage) and advanced (BCLC C stage) liver cancer patients:

  1. A single tumor > 5 cm, or multiple tumors > 3 cm.
  2. Diffuse hepatocellular carcinoma.
  3. Vascular invasion (e.g., portal vein obstruction).
  4. Extrahepatic tumor spread.
* Early-stage liver cancer (BCLC A stage):

  1. Contraindications for radiofrequency ablation (RFA).
  2. Target lesions previously treated with local therapies, including surgical resection, percutaneous ethanol injection (PEI), or liver transplantation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatocellular carcinoma (BCLC stage 0 and stage A) undergo radiofrequency ablation (RFA) treatment
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient liver reserve capacity before and after radiofrequency ablation therapy | 2 years
  Expressed as percentage of injected dose (%ID) and standardized uptake value (SUV).
  1. Correlation with patients' baseline characteristics, laboratory data, tumor characteristics
  2. Compared with ICG test
  3. Compared with computed tomography
  4. Correlation with patients' overall survival, progression free survival, objective response rate

IPD SHARING:
Plan to Share IPD: No